CLINICAL TRIAL: NCT05448794
Title: Efficacy of Ultrasound-guided Intra-Articular Hypertonic Dextrose(Prolotherapy) and Hydrodilatation for Frozen Shoulder
Brief Title: Efficacy of Prolotherapy and Hydrodilatation for Frozen Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ya Chang, MD, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C202105038 TSGHIRB
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- evaluation prolotherapy for frozen shoulder (Experimental): This pilot study highlighted that prospective studies are required to prove its clinical application for FS and other conditions.
  Interventions: Other: injection

INTERVENTIONS:
Other: injection — ultrasound-guided hydrodilatation with hypertonic Dextrose

SUMMARY:
Objective: To determine whether ultrasound-guided Intra-Articular Hypertonic Dextrose and hydrodilatation improves pain and function in patients with frozen shoulder(FS)

DETAILED DESCRIPTION:
Setting: a medical center hospital. Participants: Subjects with primary FS with shoulder pain more than 3 months. Interventions: Participants randomly be assigned into A and B group: group A received ultrasound-guided hydrodilatation with hypertonic Dextrose with a mixture of 2mL of 50%, 1mL of 2% lidocaine, and 6ml normative saline ; group B : ultrasound-guided hydrodilatation with 9 mL of normative saline and 1 mL of 2% lidocaine.

Main Outcome Measures: The primary outcome measure was the Shoulder Pain and Disability Index score. Secondary outcomes were the VAS of shoulder pain level, muscle power and angles of shoulder passive range of motion, including flexion, abduction, extension, external rotation, and internal rotation at pretreatment and weeks 2, 4, 8, 12 and 24 of post-treatment.

ELIGIBILITY:
Participants diagnosed with primary FS who had experienced shoulder pain for more than 6 months and a reduction > 30° in passive ROM of the affected shoulder in at least two directions (forward flexion, abduction, or external rotation) compared with the contralateral side were evaluated for eligibility. 23 Subjects with any degree of tear or calcified tendinitis of rotator cuff tendons, previous shoulder surgery, previous intra-articular injection for the affected shoulder within 3 months of the study; or any secondary FS caused by metabolic, rheumatic, infectious arthritis, stroke, tumor, shoulder fracture/dislocation, or acute cervical radiculopathy were excluded. 23

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-08-22 (Estimated)

PRIMARY OUTCOMES:
the Shoulder Pain and Disability Index score | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YA CHANG, MD, Study Director — Tri-Service General Hospital, School of Medicine, National Defense Medical Center, Taipei, Taiwan.
Locations (1):
- Tri-Service General Hospital, Taipei, Alberta, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
after publish, we could share our plan
Supporting Information: Study Protocol
Time Frame: after publish
Access Criteria: we will discuss our all authors